CLINICAL TRIAL: NCT00799604
Title: An Open-label Study in Patients Undergoing Cardiac Surgery to Evaluate the Effect of Bolus Clevidipine Administration (SPRINT)
Brief Title: Clevidipine Bolus Administration in the Treatment of Hypertensive Patients Undergoing Cardiac Surgery (SPRINT)
Acronym: SPRINT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMC-CLV-08-02
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Hypertension
Keywords: Hypertension; Antihypertensive Agent; Calcium Channel Blocker
MeSH Terms: conditions — Hypertension | interventions — clevidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- clevidipine (Experimental): Patients were sequentially assigned to one of following three planned dose cohorts for Bolus 1 within the clevidipine arm:
  * Cohort 1: clevidipine 250 µg (0.5 mL)
  * Cohort 2: clevidipine 500 µg (1 mL)
  * Cohort 3: clevidipine 125 µg (0.25 mL or 0.5 mL of a 1:1 solution)
  Interventions: Drug: clevidipine

INTERVENTIONS:
Drug: clevidipine — Clevidipine (0.5mg/mL in 20% lipid emulsion) was administered as an IV bolus (<5 sec) by rapid injection for Bolus 1 and for Bolus 2, if second bolus dose was administered, directly into a peripheral venous catheter followed by a normal saline flush (10mL).
  Other Names: clevidipine injectable emulsion; clevidipine emulsion; Cleviprex

SUMMARY:
This study was designed to evaluate the pharmacodynamics of a bolus dosing regimen of clevidipine, a vascular-selective L-type calcium channel antagonist, for the management of blood pressure in cardiac surgery patients, as well as to evaluate the efficacy, safety and pharmacokinetics of clevidipine after bolus administration.

DETAILED DESCRIPTION:
Study participants were screened up to 14 days prior to their elective cardiac surgery. For the purpose of this study, hypertension was defined as systolic blood pressure (SBP) ≥140 mm Hg immediately prior to initiation of study drug.

On the day of surgery, an IV bolus dose of clevidipine (Bolus 1 - pre-anesthesia) was administered to each eligible study participant during Treatment Period 1 to decrease BP before induction of general anesthesia. The dose (either 125 μg, 250 μg or 500 μg) given was based on the assigned cohort for each participant, listed in the 'Arms' section below.

At the discretion of the investigator, a second IV bolus dose of clevidipine (Bolus 2 - with anesthesia) could have been administered during Treatment Period 2 at either 125 μg, 250 μg or 500 μg, based upon the earlier observed response to Bolus 1. This dose was administered after the induction of anesthesia, to decrease BP prior to cannulation of the ascending aorta for initiation of cardiopulmonary bypass.

Assessment of safety was performed throughout Treatment Periods 1 and 2 with Adverse Events (AEs) followed 6 hours post final bolus dose and Serious Adverse Events (SAEs) followed 24 hours post final bolus dose.

ELIGIBILITY:
Inclusion Criteria:

* Require elective cardiac operation involving the use of cardiopulmonary bypass
* Age 18 years or older
* A history or hypertension and/or expected to require perioperative antihypertensive therapy in the opinion of the investigator
* Written informed consent
* Pre-anesthesia baseline SBP ≥140 mm Hg just prior to bolus, measured using an arterial line

Exclusion Criteria:

* Receiving either intravenous vasopressor or intravenous vasodilatory therapy in the 72 hours prior to dosing
* Critical left main coronary artery stenosis
* Critical aortic valve (<0.5 cm3) or mitral valve (<1.0 cm3) stenosis
* Acute myocardial infarction within the prior 14 days
* Fully paced cardiac rhythm
* Known or suspected aortic dissection
* Requiring preoperative intra-aortic balloon pump counterpulsation therapy
* Contraindication to transesophageal echocardiography
* Positive pregnancy test or breast feeding
* Intolerance or allergy to calcium channel blockers
* Allergy to soybean oil or egg lecithin
* Any condition(s) that in the Investigator's opinion would warrant exclusion from the study or prevent the patient from completing the study
* Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert T. Cheung, MD, Principal Investigator — University of Pennsylvania; Edwin G. Avery, IV, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Harvard Medical School, Boston, Massachusetts
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty patients were enrolled at two hospitals. All received an initial dose of clevidipine (Bolus 1-pre-anesthesia) during Treatment Period 1; 21 participants received a second bolus dose (Bolus 2-with anesthesia)during Treatment 2 per the discretion of the investigator at 250, 500 or 125μg, depending on patient response to Bolus 1.
Pre-assignment Details: A screening period began up to 14 days prior to study drug administration, consisting of obtaining informed consent, confirming patient eligibility, and collecting screening assessments. Patient eligibility was further verified on treatment day to confirm SPB ≥140 mm Hg prior to study drug. If SBP was <140 mm Hg, no study drug was administered.
Groups:
- Planned Cohort 1: Clevidipine 250 μg (0.5 mL): Clevidipine was administered at 250 μg during Treatment Period 1 prior to induction of general anesthesia as an IV bolus (<5 seconds) (Bolus 1 - pre-anesthesia) by rapid injection. At the discretion of the investigator, a second bolus (Bolus 2 - with anesthesia) could be administered during Treatment Period 2 after induction of general anesthesia at 125 μg, 250 μg or 500 μg based upon the earlier observed response to Bolus 1. Five participants who received a Bolus 1 dose of 250 μg during Treatment Period 1 and one participant who received a Bolus 1 dose of 125 μg during Treatment Period 1 received a Bolus 2 dose of 250 μg during Treatment Period 2 in this cohort.
- Planned Cohort 2: Clevidipine 500 μg (1.0 mL): Clevidipine was administered at 500 μg during Treatment Period 1 prior to induction of general anesthesia as an IV bolus (<5 seconds) (Bolus 1 - pre-anesthesia) by rapid injection. At the discretion of the investigator, a second bolus (Bolus 2 - with anesthesia) could be administered during Treatment Period 2 after induction of general anesthesia at 125 μg, 250 μg or 500 μg based upon the earlier observed response to Bolus 1. Six participants who received a Bolus 1 dose of 500 μg and six participants who received a Bolus 1 dose of 125 μg during Treatment Period 1 received a Bolus 2 dose of 500 μg during Treatment Period 2 in this cohort.
- Planned Cohort 3: Clevidipine 125 μg (0.25 mL or 0.5mL Sol): Clevidipine was administered at 125 μg during Treatment Period 1 prior to induction of general anesthesia as an IV bolus (<5 seconds) (Bolus 1 - pre-anesthesia) by rapid injection. At the discretion of the investigator, a second bolus (Bolus 2 - with anesthesia) could be administered during Treatment Period 2 after induction of general anesthesia at 125 μg, 250 μg or 500 μg based upon the earlier observed response to Bolus 1. Three participants who received a Bolus 1 dose of 250 μg during Treatment Period 1 received a Bolus 2 dose of 125 μg during Treatment Period 2 in this cohort.
Period: Bolus 1 (Pre-anesthesia)
Arm/Group | Planned Cohort 1: Clevidipine 250 μg (0.5 mL) | Planned Cohort 2: Clevidipine 500 μg (1.0 mL) | Planned Cohort 3: Clevidipine 125 μg (0.25 mL or 0.5mL Sol)
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0
Period: Bolus 2 (With Anesthesia)
Arm/Group | Planned Cohort 1: Clevidipine 250 μg (0.5 mL) | Planned Cohort 2: Clevidipine 500 μg (1.0 mL) | Planned Cohort 3: Clevidipine 125 μg (0.25 mL or 0.5mL Sol)
Started | 6 (Dose determined per discretion of investigator at 250, 500 or 125μg, based on response to Bolus 1.) | 12 (Dose determined per discretion of investigator at 250, 500 or 125μg, based on response to Bolus 1.) | 3 (Dose determined per discretion of investigator at 250, 500 or 125μg, based on response to Bolus 1.)
Completed | 6 | 12 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: These analyses include the Safety population defined as all participants, irrespective of eligibility, who were enrolled in Treatment Period 1 (Bolus 1 - pre-anesthesia) and were dosed with clevidipine. The number of participants in the Safety population and Modified Intent-To-Treat (mITT) population are identical.
Groups:
- Cohort 1: Clevidipine 250 μg (0.5 mL); Cohort 2: Clevidipine 500 μg (1.0 mL); Cohort 3: Clevidipine 125 μg ( mL): Baseline characteristics are reflective of the participant groupings during Treatment Period 1 (10 participants per cohort) during which clevidipine was administered at 250 μg prior to induction of general anesthesia as an IV bolus (Bolus 1 - pre-anesthesia) by rapid injection (<5 seconds).
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Clevidipine 250 μg (0.5 mL) | Cohort 2: Clevidipine 500 μg (1.0 mL) | Cohort 3: Clevidipine 125 μg ( mL) | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (11.88) | 66.4 (8.62) | 60.2 (8.85) | 62.4 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants] — These results represent Treatment Period 1 (Bolus 1 - pre-anesthesia).
  Participants
    Female | 2 | 3 | 1 | 6
    Male | 8 | 7 | 9 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — These results represent participant groupings during Treatment Period 1 (Bolus 1 - pre-anesthesia).
  Participants
    Hispanic or Latino | 0 (0) | 0 (0) | 0 (0) | 0 (0)
    Not Hispanic or Latino | 10 (100.0) | 10 (100.0) | 10 (100.0) | 30 (100.0)
    Unknown or Not Reported | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 10 | 10 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — These results represent patient groupings during Treatment Period 1 (Bolus 1 - pre-anesthesia).
  participants
    United States | 10 | 10 | 10 | 30
Height [Mean (Standard Deviation); unit: centimeters (cm)] — These results represent the participant groupings during Treatment Period 1 (Bolus 1 - pre-anesthesia).
  centimeters (cm) | 174.96 (10.381) | 168.15 (11.462) | 176.35 (9.663) | 173.15 (10.792)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] — These results represent the participant groupings during Treatment Period 1 (Bolus 1 - pre-anesthesia).
  kilograms (kg) | 81.65 (15.374) | 79.24 (12.639) | 105.05 (24.724) | 88.65 (21.279)
Screening Blood Pressure [Mean (Standard Deviation); unit: mm Hg] — These results represent the participant groupings in Treatment Period 1 (Bolus 1 - pre-anesthesia).
  mm Hg
    Systolic Blood Pressure (SBP) | 159.0 (17.45) | 170.2 (16.33) | 175.5 (19.43) | 168.2 (18.53)
    Diastolic Blood Pressure (DBP) | 80.0 (8.71) | 74.1 (10.29) | 77.7 (11.51) | 77.3 (10.18)
Screening Heart Rate [Mean (Standard Deviation); unit: Beats Per Minute (BPM)] — These results represent the participant groupings during Treatment Period 1 (Bolus 1 - pre-anesthesia).
  Beats Per Minute (BPM) | 73.1 (18.69) | 68.5 (10.42) | 69.3 (10.49) | 70.3 (13.43)

OUTCOME MEASURES:

1. Primary Outcome: The Mean Maximum Absolute Change in Systolic Blood Pressure From Baseline Within 15 Minutes From the First Bolus Dose of Clevidipine (Treatment Period 1, Bolus 1 - Pre-anesthesia).
Description: Blood Pressure was measured at 60, 45, 30, 0 seconds prior to first Bolus dose (Bolus 1), and every 5 seconds after Bolus 1 for 15 minutes. Baseline SBP of Bolus 1 is defined as, 'median of all measurements prior to or at the start of Bolus 1'. Locally weighted scatterplot smoothing (LOWESS) method was used to determine the minimum SBP value for each patient. Maximum absolute change is the minimum SBP value within 15 minutes from bolus 1 minus baseline value.
Time Frame: From start to 15 minutes of Bolus 1 dose of clevidipine (pre-anesthesia).
Population: Modified Intent-to-Treat (mITT) population: all enrolled patients who were deemed eligible for the study by meeting all inclusion and no exclusion criteria and were treated with clevidipine. The mITT population is the primary population for the analyses of efficacy.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Cohort 1: Clevidipine 250 μg (0.5 mL): Clevidipine was administered at 250 μg during Treatment Period 1 prior to induction of general anesthesia as an IV bolus (Bolus 1 - pre-anesthesia) by rapid injection (<5 seconds).
- Cohort 2: Clevidipine 500 μg (1.0 mL): Clevidipine was administered at 500 μg during Treatment Period 1 prior to induction of general anesthesia as an IV bolus (Bolus 1 - pre-anesthesia) by rapid injection (<5 seconds).
- Cohort 3: Clevidipine 125 μg (0.25 mL or 0.5 mL of a 1:1 Sol): Clevidipine was administered at 125 μg during Treatment Period 1 prior to induction of general anesthesia as an IV bolus (Bolus 1 - pre-anesthesia) by rapid injection (<5 seconds).
Arm/Group | Cohort 1: Clevidipine 250 μg (0.5 mL) | Cohort 2: Clevidipine 500 μg (1.0 mL) | Cohort 3: Clevidipine 125 μg (0.25 mL or 0.5 mL of a 1:1 Sol)
Number analyzed (Participants) | 10 | 10 | 10
mm Hg | -18.8 (6.51) | -37.0 (17.76) | -15.8 (11.43)

2. Secondary Outcome: The Percentage of Patients With Systolic Blood Pressure ≤85 mm Hg Within 15 Minutes From the First Bolus Dose of Clevidipine (Treatment Period 1, Bolus 1 - Pre-anesthesia).
Description: The percentage is calculated using the number of patients with a systolic blood pressure ≤85 mm Hg within 15 minutes from the initial Bolus 1 dose divided by the total number of patients who were treated with a Bolus 1 clevidipine, and multiplied by 100.
Time Frame: From start to 15 minutes of Bolus 1 dose of clevidipine (pre-anesthesia).
Population: Modified Intent-to-Treat (mITT) population: all enrolled patients who are eligible for the study and treated with clevidipine. The mITT population will be the primary population for the analyses of efficacy.
Measure: Number (95% Confidence Interval); unit: percent patients
Groups:
- Cohort 3: Clevidipine 125 μg (0.25 mL or 0.5 mL): Clevidipine was administered at 125 μg during Treatment Period 1 prior to induction of general anesthesia as an IV bolus (Bolus 1 - pre-anesthesia) by rapid injection (<5 seconds).
Arm/Group | Cohort 1: Clevidipine 250 μg (0.5 mL) | Cohort 2: Clevidipine 500 μg (1.0 mL) | Cohort 3: Clevidipine 125 μg (0.25 mL or 0.5 mL)
Number analyzed (Participants) | 10 | 10 | 10
percent patients | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: The Median Time to 5%, 10%, and 15% Systolic Blood Pressure Reduction From Baseline Within 15 Minutes From the First Bolus Dose of Clevidipine (Treatment Period 1, Bolus 1 -Pre-anesthesia).
Description: BP was measured at 60, 45, 30, 0 seconds prior to first Bolus dose (bolus 1), and every 5 seconds after Bolus 1 for 15 minutes. Baseline SBP of bolus 1 is defined as median of all measurements prior to or at the start of Bolus 1. The time at which first target SBP reduction (ex. 5%) from baseline was reached was identified for each patient using fitted values from LOWESS method. Kaplan-Meier method was used to estimate the median time. Patients who never reached 5%, 10% or 15% reduction, withdrew from study or changed antihypertensive within 15 minutes were censored.
Time Frame: From start to 15 minutes of Bolus 1 of clevidipine (pre-anesthesia).
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Cohort 1: Clevidipine 250 μg (0.5 mL) | Cohort 2: Clevidipine 500 μg (1.0 mL) | Cohort 3: Clevidipine 125 μg (0.25 mL or 0.5 mL)
Number analyzed (Participants) | 10 | 10 | 10
minutes
  5 % Reduction | 0.9 [0.8 to 1.4] | 0.8 [0.2 to 1.3] | 1.0 [0.7 to NA] — Not Estimable: Unable to be determined due to a lack of enough participants achieving a 5% systolic blood pressure reduction within 15 minutes within this cohort.
  10% Reduction | 1.3 [1.0 to NA] — Not Estimable: Unable to be determined due to a lack of enough participants achieving a 10% systolic blood pressure reduction within 15 minutes within this cohort. | 1.1 [0.4 to 1.3] | NA [NA to NA] — Not Estimable: Unable to be determined due to a lack of enough participants achieving a 10% systolic blood pressure reduction within 15 minutes within this cohort.
  15% Reduction | NA [NA to NA] — Not Estimable: Unable to be determined due to a lack of enough participants achieving a 15% systolic blood pressure reduction within 15 minutes within this cohort. | 1.2 [0.8 to NA] — Not Estimable: Unable to be determined due to a lack of enough participants achieving a 15% systolic blood pressure reduction within 15 minutes within this cohort. | NA [NA to NA] — Not Estimable: Unable to be determined due to a lack of enough participants achieving a 15% systolic blood pressure reduction within 15 minutes within this cohort.

4. Secondary Outcome: The Mean Percent Change in Systolic Blood Pressure From Baseline Over Time During the First 15 Minutes Following First Bolus Dose of Clevidipine (Treatment Period 1, Bolus 1 - Pre-anesthesia).
Description: BP was measured at 60, 45, 30, 0 seconds prior to first Bolus dose (Bolus 1), and every 5 seconds after Bolus 1 for 15 minutes. Baseline SBP of Bolus 1 is defined as median of all measurements prior to or at the start of Bolus 1. SBP change (percent change) from baseline is calculated at each collection time point after bolus 1 dose for each patient.
Time Frame: From start to 15 minutes of Bolus 1 of clevidipine (pre-anesthesia).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1: Clevidipine 250 μg (0.5 mL) | Cohort 2: Clevidipine 500 μg (1.0 mL) | Cohort 3: Clevidipine 125 μg (0.25 mL or 0.5 mL)
Number analyzed (Participants) | 10 | 10 | 10
percent change
  SBP 0.25 minutes after Bolus 1 | 0.96 (4.346) | -0.10 (7.585) | 0.18 (3.034)
  SBP 0.5 minutes after Bolus 1 | 2.79 (5.397) | -2.41 (6.057) | -1.59 (3.172)
  SBP 0.75 minutes after Bolus 1 | -5.22 (4.916) | -9.09 (6.901) | -5.87 (3.705)
  SBP 1 minute after Bolus 1 | -8.37 (4.181) | -12.29 (8.714) | -5.67 (5.848)
  SBP 1.5 minutes after Bolus 1 | -8.64 (3.031) | -19.40 (8.744) | -6.68 (3.694)
  SBP 2 minutes after Bolus 1 | -9.51 (4.669) | -20.36 (10.773) | -7.07 (5.336)
  SBP 3 minutes after Bolus 1 | -6.58 (5.492) | -17.95 (9.732) | -6.79 (5.665)
  SBP 5 minutes after Bolus 1 | -4.23 (4.506) | -11.08 (5.711) | -3.07 (4.170)
  SBP 7 minutes after Bolus 1 | -1.31 (4.909) | -6.77 (7.837) | -3.17 (3.443)
  SBP 15 minutes after Bolus 1 | 0.58 (6.119) | -0.33 (14.384) | -2.32 (3.347)

5. Secondary Outcome: The Median Time to 50%, and, When Available, 90% Recovery From Maximum SBP Effect Following the First Bolus Dose of Clevidipine for Patients Who Achieved the Endpoints (Treatment Period 1, Bolus 1 - Pre-anesthesia).
Description: Analysis is of the time in minutes between the recorded time at the maximum absolute change and the time of the systolic blood pressure value at the first 50% recovery. The 50% recovery value is equal to the minimum recorded systolic blood pressure value plus 50% of the maximum amount of systolic blood pressure reduction (the Bolus 1 baseline value minus the value at the maximum absolute change).
Time Frame: Up to 15 minutes following the first bolus dose of clevidipine (pre-anesthesia).
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: minutes
Groups:
- Cohort 3: Clevidipine 125 μg (0.25 mL or 0.5 mL Sol): Clevidipine was administered at 125 μg during Treatment Period 1 prior to induction of general anesthesia as an IV bolus (Bolus 1 - pre-anesthesia) by rapid injection (<5 seconds).
Arm/Group | Cohort 1: Clevidipine 250 μg (0.5 mL) | Cohort 2: Clevidipine 500 μg (1.0 mL) | Cohort 3: Clevidipine 125 μg (0.25 mL or 0.5 mL Sol)
Number analyzed (Participants) | 10 | 10 | 10
minutes
  Time to 50% recovery in SBP | 1.8 [0.4 to 3.9] | 2.9 [1.8 to 4.4] | 2.5 [1.1 to NA] — Not Estimable: Not reached since >50% of patients did not achieve 50% of recovery within 15 min.
  Time to 90% recovery in SBP | 5.2 [2.1 to NA] — Not Estimable: Not reached since >50% of patients did not achieve 90% of recovery within 15 min. | 6.8 [3.1 to NA] — Not Estimable: Not reached since >50% of patients did not achieve 90% of recovery within 15 min. | NA [NA to NA] — Not Estimable: Not reached since >50% of patients did not achieve 90% of recovery within 15 min.

6. Secondary Outcome: Change in Heart Rate After Bolus 1 (Pre-anesthesia).
Description: The baseline heart rate was measured as the median of all the heart rate measurements within 60 seconds or at the start of the administration of Bolus 1.
Time Frame: Baseline up until the first 15 minutes following Bolus 1 (pre-anesthesia).
Population: Safety population: all enrolled patients (irrespective of eligibility) who are dosed with clevidipine. The safety population will be the primary population used for the safety analyses.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Cohort 1: Clevidipine 250 μg (0.5 mL) | Cohort 2: Clevidipine 500 μg (1.0 mL) | Cohort 3: Clevidipine 125 μg (0.25 mL or 0.5 mL)
Number analyzed (Participants) | 10 | 10 | 10
beats per minute (bpm) | 11.0 (10.15) | 3.1 (2.73) | 2.0 (2.83)

7. Primary Outcome: The Mean Maximum Percent Change in Systolic Blood Pressure From Baseline Within 15 Minutes From the First Bolus Dose of Clevidipine (Treatment Period 1, Bolus 1 - Pre-anesthesia).
Description: Blood Pressure was measured at 60, 45, 30, 0 seconds prior to first Bolus dose (Bolus 1), and every 5 seconds after Bolus 1 for 15 minutes. Baseline SBP of Bolus 1 is defined as, 'median of all measurements prior to or at the start of Bolus 1'. Locally weighted scatterplot smoothing (LOWESS) method was used to determine the minimum SBP value for each patient. Maximum percent change is defined as the maximum absolute change divided by the baseline value of bolus 1 and multiplied by 100.
Time Frame: From start to 15 minutes of Bolus 1 dose of clevidipine (pre-anesthesia).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1: Clevidipine 250 μg (0.5 mL) | Cohort 2: Clevidipine 500 μg (1.0 mL) | Cohort 3: Clevidipine 125 μg (0.25 mL or 0.5 mL of a 1:1 Sol)
Number analyzed (Participants) | 10 | 10 | 10
percent change | -11.89 (3.851) | -22.10 (9.288) | -8.91 (5.966)

ADVERSE EVENTS:
Time Frame: Non-serious AE(s) were documented and assessed following initiation of clevidipine administration through 6 hours post final bolus dose. SAEs were assessed up to 24 hours post final bolus dose, regardless of causal relationship to the study drug.
Groups:
- All Participants Across All Cohorts and Treatment Periods: Study participants were sequentially assigned one of three cohorts to receive either a 250 μg, 500 μg or 125 μg bolus dose of clevidipine during Treatment Period 1 prior to induction of general anesthesia (Bolus 1 - pre-anesthesia) by rapid injection (<5 seconds). At the discretion of the investigator, a second bolus could be administered during Treatment Period 2 after induction of general anesthesia (Bolus 2 - with anesthesia) at 125 μg, 250 μg or 500 μg based upon the earlier observed response to Bolus 1.
Arm/Group | All Participants Across All Cohorts and Treatment Periods
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 12/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants Across All Cohorts and Treatment Periods (N=30)
Encephalopathy (Nervous system disorders) | 1 (1) — unrelated
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants Across All Cohorts and Treatment Periods (N=30)
Acidosis (Metabolism and nutrition disorders) | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4
Hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The site agrees that publication of Study results at the site is not permitted until after the presentation and publication of the multi-center results or an affirmative decision is made by Sponsor not to proceed with such publication. In such a case, Sponsor shall provide access to all Study site data to the academic Study Coordination Center, or upon request Sponsor will provide access to all Study site data to Institution. The site will adhere to terms for Sponsor review prior to submission.